CLINICAL TRIAL: NCT01429961
Title: Phase II Trial of Palliative Chemotherapy With TS-1 and Oxaliplatin for Patients With Advanced Hepatocellular Carcinoma
Brief Title: Trial of Palliative Chemotherapy With TS-1 and Oxaliplatin for Patients With Advanced Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-1010-054-336
Record Dates: First submitted 2011-09-06; First posted 2011-09-07 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-09

CONDITIONS: Advanced Hepatocellular Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SOX (Experimental): TS-1, Oxaliplatin regimen (3week) Oxaliplatin 130 mg/m2 IV Day 1 S-1 40 mg/m2 b.i.d. Day1-14
  Interventions: Drug: SOX

INTERVENTIONS:
Drug: SOX — TS-1, Oxaliplatin regimen (3week) Oxaliplatin 130 mg/m2 IV Day 1 S-1 40 mg/m2 b.i.d. Day1~14

SUMMARY:
Phase II trial of Palliative Chemotherapy with TS-1 and Oxaliplatin for Patients with Advanced Hepatocellular Carcinoma

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* ECOG performance score of two or less
* Child Pugh class A•
* Histologically or cytologically confirmed HCC or clinical diagnosis of HCC when the following criteria are all met History of chronic hepatitis or cirrhosis of liver Typical features of HCC demonstrated in dynamic imaging studies, such as three phase computed tomography AFP level more than 200 ng/mL
* presence of extrahepatic measurable lesion
* no prior systemic therapy (excluding sorafenib)
* adequate marrow, liver, kidney function
* written informed consent

Exclusion Criteria:

* prior systemic therapy (excluding sorafenib)
* hypersensitivity to study drugs
* active gastrointestinal bleeding
* other malignancies within five years
* pregnant or breastfeeding female
* symptomatic brain or leptomeningeal metastasis
* clinically significant heart disease
* interstitial pneumonia
* peripheral neuropathy grade one or more
* uncontrolled infection
* renal impairment
* prior use of investigational drug or therapy within 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2011-05; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Time to progression (TTP) | 2 years
  The time from study enrollment to tumor progression or death

SECONDARY OUTCOMES:
overall survival | 2 years
  overall survival
response rate | 2 years
  response rate by RECIST 1.1
toxicity | 2 years
  toxicity according to NCI-CTCAE v.3.0

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Lee DW, Lee KH, Kim HJ, Kim TY, Kim JS, Han SW, Oh DY, Kim JH, Im SA, Kim TY. A phase II trial of S-1 and oxaliplatin in patients with advanced hepatocellular carcinoma. BMC Cancer. 2018 Mar 5;18(1):252. doi: 10.1186/s12885-018-4039-9. PMID 29506478